CLINICAL TRIAL: NCT00267774
Title: Fractional Flow Reserve Versus Angiography for Multivessel Evaluation (F.A.M.E.)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, William Fearon, Principle Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3933
Record Dates: First submitted 2005-12-19; First posted 2005-12-21 (Estimated); Results first posted 2016-07-27 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-10

CONDITIONS: Coronary Arteriosclerosis
MeSH Terms: conditions — Coronary Artery Disease

ARMS (2):
- FFR guided PCI (Experimental)
  Interventions: Device: Fractional flow reserve
- Angio-guided PCI (Active Comparator)
  Interventions: Procedure: Angio-guided PCI

INTERVENTIONS:
Device: Fractional flow reserve
  Arms: FFR guided PCI
Procedure: Angio-guided PCI
  Arms: Angio-guided PCI

SUMMARY:
In this multicenter, international study we are evaluating two approaches to determine which coronary artery narrowings require stent placement in patients with multivessel coronary artery disease. Patients will be randomized to an angiographic strategy, where only coronary angiography is used to determine which lesions to stent or to a pressure wire strategy where fractional flow reserve, an index measured with the pressure wire, will be used to determine which lesions to stent. The primary outcome will be major adverse cardiac events at 1 year. A secondary outcome will be cost-effectiveness.

DETAILED DESCRIPTION:
Detailed protocol

* If a patient is eligible for the study (see inclusion and exclusion criteria) and has given informed consent, the operator has to define all lesions with a stenosis severity of at least 50% by visual estimate in which he would consider stent implantation. These stenoses are noted on a scheme of the coronary arteries before randomization.
* Thereafter, randomization is performed to the FFR-guided strategy or the angiography-guided strategy. If the patient is randomized to the angiography-guided strategy, all the lesions indicated beforehand, will be stented with drug-eluting stents. If the patient is assigned to the FFR-guided group, fractional flow reserve is measured in all lesions and only those lesions are stented with a fractional flow reserve </=0.80. Treatment after PCI is according to local routine and should include at least aspirin 80 mg daily and clopidogrel (Plavix) 75 mg per day for at least 12months.
* FFR should be determined by using i.v. adenosine 140 µg/kg/min, in order to make pull-back recordings and analyze different abnormalities along the coronary arteries. Adenosine i.v. by the femoral venous route, is mandatory for participation in the study.
* In case of serial stenosis, FFR 'of the complete vessel' should be </= 0.80 to warrant PCI of one of more of these lesions in case the patient belongs to the FFR-guided group. In case of the angio-guided group, every lesion >50% by visual estimation that the operator indicated a prior as requiring stenting, should be stented (this is mandatory). Long stents to cover a segment or multiple shorter stents, can be placed at the discretion of the operator.

Follow-up

All patients will be followed up after 1 month (±1 week), 6 months (±1 month), and 1 year (±1 month). All adverse cardiac events (death, acute MI, CABG or [re]-PCI will be noted, as well as functional class and number of anti-anginal drugs. If a patient is admitted to a hospital because of an acute coronary syndrome, repeat angiography is strongly advocated to define if the event is related to one of the deferred lesions or to one of the non-deferred lesions. If the patient belongs to the FFR-guided arm, repeat measurement of FFR is advocated for all lesions. If, during follow-up, patients in the FFR-guided group have to undergo coronary angiography because of recurrent angina or any other reason without an event, pressure measurement should be repeated as well.

On the contrary, once a patient has been assigned to the angiographic guided group, this strategy should be followed consistently during follow-up investigations. For example, if a patient in the angiographic guided arm has recurrent chest pain, undergoes angiography, and is found to have in-stent restenosis, re-PCI should be performed based on the angiogram and pressure wire use is prohibited.

In other words, the strategy to which the patient has been assigned initially, should be followed during the entire study period.

Endpoints

Primary endpoints

1. The primary clinical endpoint is the 12-month binary major adverse cardiac event (MACE) rate. MACE is defined as:

* All cause death,
* Documented myocardial infarction,
* Repeat revascularization (PCI and/or CABG) as adjudicated by the Clinical Event Committee

Secondary endpoints

1. Global cost effectiveness after one year
2. Cardiac death and myocardial infarction rate at 1 year
3. Functional class at 1 year.
4. Number of anti-anginal drugs after 1 year
5. Overall MACE rate at 1 month post-procedure and at 6 months, 2, 3 and 5 years.
6. A comparison of outcomes based on type of drug-eluting stent.
7. Prognostic value of FFR after stenting.
8. Correlation between FFR and nuclear perfusion imaging.

ELIGIBILITY:
Inclusion Criteria:- at least 2 coronary lesions of 50% stenosis or greater in at least 2 major epicardial arteries

* age>/=18

Exclusion Criteria:-- STEMI < 5 days ago or non-STEMI with CK > 1000 U/l < 5 days ago

* Pregnancy
* Extremely tortuous or calcified coronary arteries, or other technical conditions interfering with reliable coronary pressure measurement
* Serious concomitant disease, decreasing life expectancy to <2 years
* Previous coronary bypass surgery (CABG)
* Contraindication for drug-eluting stent
* Cardiogenic shock
* Inability to give informed consent
* Suspicion of significant left main (LM) stenosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1005 (Actual)
Dates: Start 2006-01; Primary Completion 2008-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nico H Pijls, Principal Investigator — Catharina Ziekenhuis Eindhoven; William F Fearon, Principal Investigator — Stanford University
Locations (2):
- Stanford University School of Medicine, Stanford, California, United States
- Catharina Hospital, Eindhoven, Netherlands

REFERENCES:
- [Result] Fearon WF, Bornschein B, Tonino PA, Gothe RM, Bruyne BD, Pijls NH, Siebert U; Fractional Flow Reserve Versus Angiography for Multivessel Evaluation (FAME) Study Investigators. Economic evaluation of fractional flow reserve-guided percutaneous coronary intervention in patients with multivessel disease. Circulation. 2010 Dec 14;122(24):2545-50. doi: 10.1161/CIRCULATIONAHA.109.925396. Epub 2010 Nov 29. PMID 21126973
- [Result] Tonino PA, De Bruyne B, Pijls NH, Siebert U, Ikeno F, van' t Veer M, Klauss V, Manoharan G, Engstrom T, Oldroyd KG, Ver Lee PN, MacCarthy PA, Fearon WF; FAME Study Investigators. Fractional flow reserve versus angiography for guiding percutaneous coronary intervention. N Engl J Med. 2009 Jan 15;360(3):213-24. doi: 10.1056/NEJMoa0807611. PMID 19144937
- [Derived] Nishi T, Piroth Z, De Bruyne B, Jagic N, Mobius-Winkler S, Kobayashi Y, Derimay F, Fournier S, Barbato E, Tonino P, Juni P, Pijls NHJ, Fearon WF. Fractional Flow Reserve and Quality-of-Life Improvement After Percutaneous Coronary Intervention in Patients With Stable Coronary Artery Disease. Circulation. 2018 Oct 23;138(17):1797-1804. doi: 10.1161/CIRCULATIONAHA.118.035263. PMID 30354650
- [Derived] Kobayashi Y, Nam CW, Tonino PA, Kimura T, De Bruyne B, Pijls NH, Fearon WF; FAME Study Investigators. The Prognostic Value of Residual Coronary Stenoses After Functionally Complete Revascularization. J Am Coll Cardiol. 2016 Apr 12;67(14):1701-11. doi: 10.1016/j.jacc.2016.01.056. PMID 27056776
- [Derived] van Nunen LX, Zimmermann FM, Tonino PA, Barbato E, Baumbach A, Engstrom T, Klauss V, MacCarthy PA, Manoharan G, Oldroyd KG, Ver Lee PN, Van't Veer M, Fearon WF, De Bruyne B, Pijls NH; FAME Study Investigators. Fractional flow reserve versus angiography for guidance of PCI in patients with multivessel coronary artery disease (FAME): 5-year follow-up of a randomised controlled trial. Lancet. 2015 Nov 7;386(10006):1853-60. doi: 10.1016/S0140-6736(15)00057-4. Epub 2015 Aug 30. PMID 26333474
- [Derived] Nam CW, Mangiacapra F, Entjes R, Chung IS, Sels JW, Tonino PA, De Bruyne B, Pijls NH, Fearon WF; FAME Study Investigators. Functional SYNTAX score for risk assessment in multivessel coronary artery disease. J Am Coll Cardiol. 2011 Sep 13;58(12):1211-8. doi: 10.1016/j.jacc.2011.06.020. PMID 21903052
- [Derived] Pijls NH, Fearon WF, Tonino PA, Siebert U, Ikeno F, Bornschein B, van't Veer M, Klauss V, Manoharan G, Engstrom T, Oldroyd KG, Ver Lee PN, MacCarthy PA, De Bruyne B; FAME Study Investigators. Fractional flow reserve versus angiography for guiding percutaneous coronary intervention in patients with multivessel coronary artery disease: 2-year follow-up of the FAME (Fractional Flow Reserve Versus Angiography for Multivessel Evaluation) study. J Am Coll Cardiol. 2010 Jul 13;56(3):177-84. doi: 10.1016/j.jacc.2010.04.012. Epub 2010 May 28. PMID 20537493

RESULTS

PARTICIPANT FLOW:
Groups:
- FFR Guided PCI: Fractional flow reserve
- Angio-guided PCI: Angio-guided PCI
Period: Overall Study
Arm/Group | FFR Guided PCI | Angio-guided PCI
Started | 509 | 496
Completed | 509 | 496
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FFR Guided PCI | Angio-guided PCI | Total
Number analyzed (Participants) | 509 | 496 | 1005
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (10.3) | 64.2 (10.2) | 64.4 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125 | 136 | 261
  Male | 384 | 360 | 744

OUTCOME MEASURES:

1. Primary Outcome: Major Adverse Cardiac Events
Description: All cause death, Documented myocardial infarction, Repeat revascularization (PCI and/or CABG) as adjudicated by the Clinical Event Committee
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | FFR Guided PCI | Angio-guided PCI
Number analyzed (Participants) | 509 | 496
participants | 67 | 91

2. Secondary Outcome: Cost Effectiveness Measured as Index Procedural and Hospitalization Costs
Description: Costs for each strategy included the initial procedural costs and costs during the 1-year follow-up. The costs of the index procedures were calculated from the actual resource consumption by determining the amount of guiding catheters, regular wires, pressure wires, balloon dilatation catheters, stents, antiplatelet therapy, adenosine, contrast media, and hospital days used for each patient's index procedure. These were multiplied by the cost of each resource in US dollars. All costs were converted to 2008 US dollars using the consumer price index (www.bls.gov).
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: US dollars
Arm/Group | FFR Guided PCI | Angio-guided PCI
Number analyzed (Participants) | 509 | 496
US dollars | 13,182 (9667) | 14,878 (9509)
Statistical Analysis 1: Comparison: FFR Guided PCI vs Angio-guided PCI; Test type: Other; p < 0.0001, t-test, 2 sided — A 2-sided value of P<0.05 was considered to indicate statistical significance

ADVERSE EVENTS:
Time Frame: 1 year
Description: Per protocol, major cardiac events were collected as adverse events.
Arm/Group | FFR Guided PCI | Angio-guided PCI
Serious Adverse Events (participants affected / at risk) | 67/509 | 91/496
Other Adverse Events (participants affected / at risk) | 0/509 | 0/496
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FFR Guided PCI (N=509) | Angio-guided PCI (N=496)
Death (Cardiac disorders) | 9 | 15
Myocardial infarction (Cardiac disorders) | 29 | 43
Repeat vascularization (Cardiac disorders) | 33 | 47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No